CLINICAL TRIAL: NCT06240130
Title: Outcome Following Use of NaOCl and Chlorhexidine as Wound Lavage Agents During Partial Pulpotomy in Mature Permanent Teeth With Symptomatic Irreversible Pulpitis: A Randomized Clinical Trial
Brief Title: Outcome Following Use of NaOCl and Chlorhexidine as Wound Lavage Agents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soumyashree Mishra
Record Dates: First submitted 2024-01-13; First posted 2024-02-02 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Irreversible Pulpitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium hypochlorite lavage group (Active Comparator): 3% sodium hypochlorite lavage will be done after pulp amputation
  Interventions: Procedure: Partial pulpotomy
- Chlorhexidine lavage group (Experimental): 2% Chlorhexidine lavage will be done after pulp amputation
  Interventions: Procedure: Partial pulpotomy

INTERVENTIONS:
Procedure: Partial pulpotomy — after caries removal and pulp exposure pulp tissue is amputated and wound lavage done with 3% NaOCl in partial pulpotomy
  Arms: Sodium hypochlorite lavage group
Procedure: Partial pulpotomy — after caries removal and pulp exposure pulp tissue is amputated and wound lavage done with 2% Chlorhexidine in partial pulpotomy
  Arms: Chlorhexidine lavage group

SUMMARY:
The goal of this clinical trial is to to compare effect of wound lavage agents NaOCl and Chlorhexidine on the outcome of partial pulpotomy in mature permanent posterior teeth with signs and symptoms indicative of irreversible pulpitis in.

The main question it aims to answer are:

Does wound lavage using chlorhexidine have equal effect as NaOCl on the outcome of partial pulpotomy in mature permanent mandibular posterior teeth with clinical signs of irreversible pulpitis?

Participants will of age group 18 to 45 years will be included and divided into two groups:

Pulp wound lavage in partial pulpotomy using 3% NaOCl as control and using 2% Chlorhexidine as experiment

DETAILED DESCRIPTION:
Title- Outcome following use of NaOCl and chlorhexidine as wound lavage agents during partial pulpotomy in mature permanent teeth with symptomatic irreversible pulpitis: A randomized clinical trial Research Question Does wound lavage using chlorhexidine have equal effect as NaOCl on the outcome of partial pulpotomy in mature permanent mandibular posterior teeth with clinical signs of irreversible pulpitis? PICO

* P (Population) - Mature permanent posterior teeth with clinical signs of symptomatic irreversible pulpitis
* I (Intervention) - 2% Chlorhexidine lavage during Partial pulpotomy
* C (Comparison) - 3% Sodium hypochlorite lavage during Partial pulpotomy
* O (Outcome) -Assessment of clinical and radiographic success at 12 months follow up To evaluate reduction in post operative pain experience at every 24 hours till 1 week
* T (time frame)- 18 months Aim-The aim of the study is to compare effect of wound lavage agents NaOCl and Chlorhexidine on the outcome of partial pulpotomy in mature permanent posterior teeth with signs and symptoms indicative of irreversible pulpitis.

Objective- Primary objective- To evaluate the clinical and radiographic success of partial pulpotomy using NaOCl or chlorhexidine as wound lavage agents in mature permanent posterior teeth with clinical signs and symptoms of irreversible pulpitis.

Secondary objective- To assess postoperative pain after partial pulpotomy using NaOCl or chlorhexidine wound lavage.

Setting: Dept. Of Conservative Dentistry & Endodontics, PGIDS, Rohtak. FINER F (feasible)= Adequate number of subjects for sample size and technical expertise are available to conduct the study I (Interesting)= The study aims to compare the effect of lavage agents (NaOCl and Chlorhexidine) on the outcome of partial pulpotomy in patients diagnosed with symptomatic irreversible pulpitis N(Novel)= No clinical trial study has compared the effect of wound lavage agents on the outcome of partial pulpotomy in mature permanent mandibular posterior teeth E(Ethical)= Ethical issues have been taken care of during the planning of the study. Subjects will be provided with information sheet and consent form. Once the study is approved by the ethical committee of the institution, it will be conducted and followed up R (Relevant)= This study will help formulate evidence-based guidelines for use of different lavage agents during partial pulpotomy in mature permanent mandibular posterior teeth.

S= Specific- yes M= Measurable- yes A= Achievable- yes R= Relevant- yes T= Time frame- 18 months

Study subjects:

Subjects of age group 18 to 45 years will be included and divided into two groups:

Pulp wound lavage in partial pulpotomy using 3% NaOCl as control and using 2% Chlorhexidine as experiment Inclusion Criteria 1) Mature permanent mandibular posterior teeth with extreme deep caries and clinical diagnosis of symptomatic irreversible pulpitis 2) Patients having normal periapical status with periapical index (PAI) score ≤ 2 and periodontally healthy teeth 3) Patients having physical status of class 1 or 2 according to ASA classification 4) Pulpal bleeding can be controlled within 10 minutes Exclusion Criteria

1. Necrotic pulp upon exposure
2. Presence of sinus tract or soft tissue swelling
3. Pregnant patients
4. Radiographic signs of internal or external root resorption Sample Size The current study is planned as an equivalent study and sample size calculated using website software www.sealedenvelope.com, which revealed that a minimum of 39 participants will be required in each group. Considering 20% loss to follow up, 49 patients will be included per group.

Randomisation Study subjects will be stratified according to age and will be randomly allocated in equal proportion to either 3% NaOCl lavage or 2% Chlorhexidine lavage group using concealed envelopes to know whether the subject would receive NaOCl rinse or Chlorhexidine rinse.

PROCEDURE After pulp exposure, amputation of superficial pulpal tissue to a depth of 2-3 mm will be done using a sterile round bur in the high-speed handpiece.

The pulp wound will be irrigated

with 3% NaOCl in with 2% Chlorhexidine in control group experimental group

Haemostasis will be achieved by placing the cotton pellet soaked with 3% NaOCl and 2% chlorhexidine in respective groups

In both groups, MTA will be and will be placed to a thickness of 2-3 mm and a layer of RMGI liner will be placed over the MTA. Then the tooth will be permanently restored with composite resin followed by immediate post operative radiograph

FOLLOW UP Patient will be recalled after 1 week, 3 months, 6 months and 1 year for clinical evaluation. Radiographic evaluation will be done after 6 months and 1 year using the same digital imaging system with standard exposure parameters as used during immediate postoperative radiograph.

Outcome Measures Primary outcome- Clinical and radiographic success rate Secondary outcome- postoperative pain experience Pain Assessment Visual analogue scale (VAS) from 0 to 100 will be used to record preoperative and post -operative pain.

Clinical Success Criteria

1. Absence of signs and symptoms of spontaneous pain or pain on stimulus and discomfort, soft tissue swelling, sinus or fistula
2. No tenderness to palpation or percussion and no periodontal probing depth
3. Positive response on EPT and cold testing Radiographic Success Criteria

1) Periapical Index (PAI) score ≤ 2 according to Orstavick 2) Absence of internal or external root resorption Statistical analysis Statistical analysis will be done using suitable statistical method

ELIGIBILITY:
Inclusion Criteria:

* Mature permanent mandibular posterior teeth with extreme deep caries and clinical diagnosis of symptomatic irreversible pulpitis
* Patients having normal periapical status with periapical index (PAI) score ≤ 2 and periodontally healthy teeth
* Patients having physical status of class 1 or 2 according to ASA classification
* Pulpal bleeding can be controlled within 10 minutes

Exclusion Criteria:

* Necrotic pulp upon exposure
* Presence of sinus tract or soft tissue swelling Pregnant patients Radiographic signs of internal or external root resorption

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Clinical Success and Radiographic Success | Base line to 12 months
  CLINICAL SUCCESS CRITERIA:
  Absence of spontaneous pain, discomfort, swelling, sinus tract or tenderness to palpation or percussion.
  RADIOGRAPHIC SUCCESS CRITERIA:
  No pathosis evident on the radiograph such as root resorption, furcal pathosis or new periapical pathosis.
  Periapical Index score 1 or 2 according to Orstavic et al.
  Evaluation of both clinical and radiographic outcome is must for analyzing the actual success of therapeutic technique. Number of participants fulfilling both clinical as well as radiographic success criteria will be considered in success category.

SECONDARY OUTCOMES:
Post operative pain | Base line to 7 days
  To assess incidence and intensity of pain postoperatively at every 24 hours till 7 days using Visual analogue Scale of 0 to 100 millimeter line. Score 0 means no pain and Score 100 means maximum pain To assess incidence and intensity of pain postoperatively at every 24 hours till 7 days using Visual analogue Scale of 0 to 100 millimeter line. Score 0 means no pain and Score 100 means maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: DR. Sanjay Tewari, MDS, Study Director — PGIDS,Rohtak, Haryana, 124001
Locations (1):
- PGIDS, Rohtak, Haryana, India

REFERENCES:
- [Derived] Mishra S, Sangwan P, Duhan J, Arora M, Mittal S, Kumar V, Ramani A. Outcome of Partial Pulpotomy in Mature Permanent Molars After Lavage With Chlorhexidine or Sodium Hypochlorite: A Randomised Clinical Trial. Int Endod J. 2026 Jan;59(1):80-90. doi: 10.1111/iej.70043. Epub 2025 Sep 30. PMID 41026352